CLINICAL TRIAL: NCT00188773
Title: Mechanism of Fatty Acid-Induced Impairment of Glucose-Stimulated Insulin Secretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Gary Lewis, University Health Network
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 03-0871-A; CDA Grant 777508221
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2007-06

CONDITIONS: Insulin Resistance Syndrome X; Pancreatic Beta Cell Function
Keywords: n-acetylcysteine,; free fatty acid,; glucose stimulated insulin secretion,; insulin resistance syndrome; antioxidant therapy; Insulin Resistance
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Acetylcysteine; soybean oil, phospholipid emulsion; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: N-acetylcysteine, intralipid, heparin — One visit subject will receive N-acetylcysteine plus intralipid and heparin, another visit n-acetylcyksteine plus saline, another visit intralipid and heparin and another visit saline alone

SUMMARY:
A prolonged elevation of plasma free fatty acids (FFA) impairs glucose stimulated insulin secretion. The concept of fatty acid impairment of glucose stimulated insulin secretion (lipotoxicity) has now been well accepted. Increased free fatty acid flux from adipose tissue to non-adipose tissue, resulting from abnormalities of fat metabolism, participates in and amplifies many of the metabolic derangements that are characteristic of insulin resistance syndrome and type 2 diabetes.

Lipotoxicity is also likely to play an important role in the progression from normal glucose tolerance to fasting hyperglycemia and conversion to frank type 2 diabetes in insulin resistant individuals. This area of research is now focused on determining the mechanisms whereby FFAs impair b-cell function. There is some evidence to suggest that lipotoxicity could be mediated through induction of reactive oxygen species (ROS). N-acetylcysteine (NAC) is a known potent antioxidant and has been used experimentally in a number of medical conditions in humans for its protective antioxidant effects. The investigators now plan to administer NAC orally to humans for 48 hours to examine the effects of antioxidant therapy in ameliorating the deleterious effects of FFAs on pancreatic beta cell function. NAC is currently approved for the treatment of acetaminophen overdose and is also used as a mucolytic agent. The investigators are now using NAC as an antioxidant to determine whether it protects the pancreatic beta cell against the toxic effects of FFAs, as outlined in the detailed study protocol. This is a proof-of-principle study and is not designed to develop n-acetylcysteine for therapeutic use.

DETAILED DESCRIPTION:
Free fatty acids will be elevated approximately 2-fold for 48 hours by intravenous infusion of Intralipid and heparin. 15 abdominally obese insulin resistant, but otherwise healthy, non-diabetic men will be studied on three occasions each, in random order, 4 weeks apart. We have chosen to study abdominally obese, insulin resistant individuals rather than lean healthy controls because we have previously shown that these individuals are more susceptible to lipotoxicity and we are therefore more likely to see differences between the interventions if differences indeed exist. Informed written consent will be obtained from all participants in accordance with the guidelines of the Human Subjects Review Committee of the University Health Network.

Subjects will be hospitalized in the Metabolic Investigation Unit (MIU) of the Toronto General Hospital for each of their three studies, which will be performed in random order 4 to 6 weeks apart. On one occasion a saline control study will be performed, on a second occasion Intralipid (20% solution @ 40ml/hr) and heparin (250u/hr) will be infused for 48 hours as previously described and on a third occasion NAC will be administered orally concurrently with the Intralipid and heparin. The dose of NAC will be the same as that recommended for acetaminophen overdose. An initial loading dose of 140mg/kg NAC followed by a maintenance dose of 70mg/kg every 4 hours during the 48 hour infusion of Intralipid and heparin. On day three, testing of glucose-stimulated insulin secretion (GSIS) will occur as outlined below. Subjects will be provided with an isocaloric diet consisting of 50% calories derived from carbohydrates, 30% fat and 20% protein during the 48 hour infusions and will fast from midnight for the testing of pancreatic beta cell function on day three.

ELIGIBILITY:
Inclusion Criteria:

The following criteria will be used for the selection of insulin resistant non-diabetic men aged 35-65 years:

1. Written informed consent obtained
2. Body mass index (BMI) > 27 kg/m2
3. Fasting triglycerides > 2 mmol/l and < 5 mmol/l
4. Waist circumference > 90 cm
5. Fasting blood glucose < 7 mmol/l
6. In order to keep the number of study subjects to a minimum (n=15), in view of the cost of these labor-intensive metabolic studies, the investigators will be studying males only 35 to 65 years of age. This will allow them to study as homogeneous a group of subjects as possible. If significant protective effects of NAC on beta cell function are detected, they will study women using a similar protocol at a later stage.
7. Hemoglobin above 130 g/L

Exclusion Criteria:

1. Patient has a history of hepatitis/hepatic disease that has been active within the previous two years
2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL) genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 100 or systolic > 180) or proliferative retinopathy
3. Fasting blood glucose > 7 mmol/l or known diabetes
4. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmias or conduction delays on ECG, unstable angina, or decompensated heart failure
5. Any laboratory values: AST > 2x ULN; ALT > 2x ULN TSH > 6 mU/l
6. Known or suspected allergy to the medication or a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reactions
7. Current addiction to alcohol or substances of abuse as determined by the investigator
8. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
9. Any lipid lowering or hypoglycemic agents
10. Previous history of asthma
11. Will not donate blood three months prior to and three months post study procedures

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-08 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To determine whether the FFA-induced impairment of pancreatic b-cell function can be ameliorated or prevented by administration of the antioxidant, NAC | 2 years
Assessment of insulin sensitivity | 2 years
To determine whether administration of NAC, an antioxidant, prevents FFA-mediated impairment of GSIS in healthy humans. | 2 years

SECONDARY OUTCOMES:
assessment of glucose stimulated insulin secretion | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary F. Lewis, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada